CLINICAL TRIAL: NCT03467321
Title: Assistant Professor, Physioterapist, PhD
Brief Title: Balance, Pulmonary Function, and Low Back Pain in Pregnant and Non-pregnant Women
Status: Completed | Type: Observational
Sponsor: Seyda TOPRAK CELENAY (Other)
Responsible Party: Sponsor-Investigator, Seyda TOPRAK CELENAY, Asist. Prof, PT, PhD, Ataturk Training and Research Hospital
Organization: Ataturk Training and Research Hospital (Other)
Other Study IDs: 2017/176
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant group: Balance with the one leg balance test with the eyes open and closed, pulmonary functions with a spirometer, and LBP with the Visual Analogue Scale (VAS) were assessed.
  Interventions: Other: Physical characteristic assessment
- Non-pregnant group: Balance with the one leg balance test with the eyes open and closed, pulmonary functions with a spirometer, and LBP with the Visual Analogue Scale (VAS) were assessed.
  Interventions: Other: Physical characteristic assessment

INTERVENTIONS:
Other: Physical characteristic assessment — Physical characteristics related to balance, pulmonary function and low back pain were evaluated

SUMMARY:
The aims of this study were to investigate balance and pulmonary functions in pregnant and non-pregnant women and to determine their relationship with LBP.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women (in the second and third trimester), non-pregnant women, aged between 18 and 40 years, volunteering to participate in the study

Exclusion Criteria:

* Having a high-risk pregnancy, preeclampsia, multiple pregnancies, gestational diabetes mellitus, hypertension, any physical disability, prior history of surgery related to spine or abdominal, spinal deformity, serious neurological, rheumatologic, cardiopulmonary or psychiatric diseases, malignancy, fracture history, or those having any exercise program or sportive activity in the last 3 months for pregnant women
* Having any physical disability, spinal or abdominal surgery, spinal deformity, serious neurological, rheumatologic, cardiopulmonary or psychiatric diseases, malignancy, or fracture history, or those having any exercise program or sportive activity in the last 3 months for non-pregnant women

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant and non pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Balance | through study completion, an average of 6 months
  Balance with the one leg balance test was assessed

SECONDARY OUTCOMES:
Pulmonary function | through study completion, an average of 6 months
  Pulmonary function with a spirometer was assessed
Low back pain | through study completion, an average of 6 months
  Low back pain with the Visual Analogue Scale was assessed

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Study Director — Ankara Yildirim Beyazıt University; Yasemin Karaaslan, Principal Investigator — Beykent University; Mete Gurol Ugur, Principal Investigator — University of Gaziantep
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)